CLINICAL TRIAL: NCT01428986
Title: Safety Study of Maraviroc's Effect on Human Osteoclasts
Acronym: MVC-Bone
Status: Completed | Type: Observational
Sponsor: National Center for Global Health and Medicine, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: FWA00005823-MVCBone2009; UMIN000006266 (Other: University hospital Medical Information Network (UMIN))
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: HIV Infections; AIDS
Keywords: maraviroc; osteoclasts; Receptors, CCR5; Chemokine CCL5
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Diabetes Mellitus, Insulin-Dependent, 22 | interventions — Maraviroc

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum, blood plasma, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Maraviroc: Those whose take maraviroc as a part of their HIV treatment
  Interventions: Drug: Maraviroc
- No maraviroc: Those who do not take maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc, 300mg BID for 72 weeks, except for cases with Efavirenz or Etravirine, 600mg BID for 72 weeks
  Other Names: Selzentry, or Celsentri
  Groups: Maraviroc

SUMMARY:
This study is to investigate the safety of maraviroc by examining whether there is bone metabolism dysfunction in actual use of maraviroc in human body, or not, measuring bone mineral density and markers for bone formation, desorption and chemokine.

DETAILED DESCRIPTION:
An observational study to investigate the safety of maraviroc by examining whether there is bone metabolism dysfunction in actual use of maraviroc in human body, or not, measuring bone mineral density and markers for bone formation, desorption and chemokine.

ELIGIBILITY:
Inclusion Criteria: Outpatients or inpatients that are treated for HIV infection at AIDS Clinical Center of National Center for Global Health and Medicine who meet all criteria following:

* Those whose primary care physician acknowledged the necessity of maraviroc treatment due to multi-resistance HIV strain that is confirmed to have CCR5 tropism.
* Those who are willing and able to consent to this study
* 20 years old or older

Exclusion Criteria: Cases applicable to ANY condition of the following:

* Those who are not suited for maraviroc (whose HIV strain to be CXCR4 tropism)
* Others who the principle investigator physician considered to be excluded

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Treatment group: primary care clinic, Non-treatment group: primary care clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of maraviroc's effect to bone metabolism and bone mineral density | 78 weeks
  Follow up HIV infected patients who take maraviroc for their bone mineral density by DEXA and for following blood/urine markers of bone metabolism and chemokine for 72 weeks:
  * Bone and chemokine markers (DPD, NTX, CTX, TRACP, BAP, osteocalcin, MIP-1alpha, MIP-1beta and RANTES)
  * Dual-energy X-ray absorptiometry

SECONDARY OUTCOMES:
Duration of the treatment efficacy | 72 weeks
  Evaluate overall HIV management status over time with:
  * Other infections: HBV, HCV, RPR, TPHA
  * HIV treatment markers: CD4, CD8, CD4/CD8, HIV-RNA
  * HAART regimens and start dates
  * Other medications: antibiotics, anticoagulants, antiplatelets, NSAID, steroids
  * Past medical history
  * HIV risk behaviors, age, sex

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Yamamoto, MD PhD, Principal Investigator — Vice Director-General of Research Institute
Locations (1):
- National Center for Global Health and Medicine, Shinjuku, Tokyo, Japan